CLINICAL TRIAL: NCT00595387
Title: Cognitive-Behavior Therapy for Bipolar Disorder
Brief Title: Effectiveness of Cognitive Behavioral Therapy for Treating Depression in People With Bipolar I Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Thilo Deckersbach, PhD, Assistant Professor Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006P001521; K23MH074895 (NIH); DSIR 83-ATP
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Bipolar Disorder; Depression
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Participants receiving supportive psychotherapy
  Interventions: Other: Supportive Psychotherapy
- 2 (Experimental): Participants receiving cognitive behavioral therapy
  Interventions: Other: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Other: Supportive Psychotherapy — Participants will attend 18 supportive therapy sessions over 5 months. Supportive psychotherapy focuses on reflecting and expressing feelings about current life issues. Participants are supported and comforted when coping with difficult situations, depression, mood swings, or anger.
  Arms: 1
Other: Cognitive Behavioral Therapy (CBT) — Participants will attend 18 CBT sessions over 5 months. CBT for depression targets depressive symptoms through a range of different treatments. This includes psychoeducation about the disorder and educating patients about the role of thoughts and behaviors in the maintenance of depressed mood. CBT also includes mood and activity monitoring, activity scheduling, and teaching participants to critically investigate and challenge negative thoughts and core beliefs that help to maintain depression.
  Arms: 2

SUMMARY:
This study will compare the effectiveness of cognitive behavioral therapy versus supportive psychotherapy in decreasing depression in people with bipolar disorder.

DETAILED DESCRIPTION:
Bipolar I disorder (BP-I) is a chronic debilitating disorder with recurrent depressive and/or manic mood episodes. Although episodes of mania are often considered the most distinguishing feature of bipolar disorder, recurrent episodes of depression make up the most functionally debilitating aspect for many individuals with BP-I. Symptoms of depressive episodes include depressed mood, lack of interest, decreased energy, low self-esteem, trouble sleeping, and change in appetite. Mood stabilizers are usually the first line of treatment for patients with bipolar disorder who are in a depressive episode, but previous research has shown that these treatments fail to bring most patients to sustained remission. As an adjunct to medication, a psychosocial treatment known as cognitive behavioral therapy (CBT) may be a promising treatment for improving depressive symptoms and for long-term stabilization in individuals with BP-I. This study will compare the effectiveness of CBT versus supportive psychotherapy in decreasing depression in people with BP-I. Using magnetic resonance imaging (MRI), this study will also assess the impact of episodic memory impairment in people with BP-I on the success of CBT treatment.

Participation in this single-blind study will last about 9 months and will include 22 study visits. There will be four pretreatment visits, during which participants will undergo a variety of tests and procedures, including interviews and questionnaires about depression and anxiety; tests on memory, attention, reaction time, and reading; and an MRI scan. Following completion of the initial assessments, participants will be randomly assigned to receive CBT or supportive psychotherapy. Participants in both groups will attend eighteen 1-hour treatment sessions over 5 months. Participants attending CBT sessions will learn specific thought processing and behavioral exercises to help reduce depressive symptoms. Participants attending psychosocial therapy sessions will learn about signs and symptoms related to depression and will be provided support in coping with their depression.

All participants will be asked to complete Mood and Memory Questionnaires before and after the first seven treatment sessions. Psychological evaluations will occur after Visits 8 and 18 of treatment and will involve the completion of questionnaires. Participants in both groups will attend a follow-up visit to evaluate tic symptoms, anxiety, and mood 4 months after the final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision (tested by vision charts)
* Diagnosis of bipolar I disorder by the Mini International Neuropsychiatric Interview (MINI)
* HAM-D score of 17 or higher

Exclusion Criteria:

* Meets criteria for DSM-IV bipolar I disorder subtype rapid cycling
* Meets criteria for DSM-IV mixed episode
* Pregnant
* Serious medical illness
* Neurologic disorder and/or head trauma
* Current or past history of selected DSM-IV Axis I disorders other than bipolar disorder, including organic mental disorder, schizophrenia, delusional disorder, and psychotic disorders not otherwise specified
* Substance abuse or dependence within the 12 months prior to study entry and/or history of substance abuse for more than 12 months
* IQ of less than 80 on the Wechsler Adult Reading Test
* Previous treatment with CBT for depression
* Contraindications to MRI (e.g., metallic implants, claustrophobia)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | Measured at baseline and Weeks 9, 20, and 36

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Deckersbach, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Bipolar Clinic and Research Program, Boston, Massachusetts, United States